CLINICAL TRIAL: NCT04646005
Title: A Phase 2 Study of Cemiplimab, an Anti-PD-1 Monoclonal Antibody, and ISA101b Vaccine in Patients With Recurrent/Metastatic HPV16 Cervical Cancer Who Have Experienced Disease Progression After First Line Chemotherapy
Brief Title: Cemiplimab and ISA101b Vaccine in Adult Participants With Recurrent/Metastatic Human Papillomavirus (HPV)16 Cervical Cancer Who Have Experienced Disease Progression After First Line Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: ISA Pharmaceuticals B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-ISA-1981; 2020-001239-29 (EudraCT Number)
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer
Keywords: HPV16 positive; Squamous histology; Recurrent; Metastatic; Adenocarcinoma/adenosquamous histology
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence; Neoplasm Metastasis; Adenocarcinoma | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cemiplimab+ISA101b (Experimental)
  Interventions: Drug: Cemiplimab; Biological: ISA101b

INTERVENTIONS:
Drug: Cemiplimab — Administered intravenously (IV) every three weeks (Q3W)
  Other Names: REGN2810; Libtayo
Biological: ISA101b — Administered by subcutaneous (SC) injection on day 1, day 29, and day 50

SUMMARY:
The primary objective of the study is to estimate the clinical benefit of cemiplimab + ISA101b after progression on first line chemotherapy, as assessed by objective response rate (ORR).

The secondary objectives of the study are:

* To characterize the safety profile of cemiplimab + ISA101b
* To assess preliminary efficacy of cemiplimab + ISA101b as measured by duration of response (DOR), progression-free survival (PFS), and overall survival (OS)

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult patients ≥18 years of age (or the legal age of adults to consent to participate in a clinical study per country specific regulations).
2. Has histologically confirmed recurrent or metastatic HPV16 positive cervical cancer as determined by an investigational HPV16 PCR assay, who have experienced disease progression after treatment with platinum containing therapy as defined in the protocol
3. Patient must be determined to be positive for HPV16 genotype, as determined by a specified central reference laboratory.
4. Patient must have measurable disease as defined by RECIST 1.1.
5. Must have received prior bevacizumab and taxol unless meets pre-specified protocol criteria
6. ECOG performance status of 0 or 1.
7. Has adequate organ and bone marrow function as defined in the protocol.
8. Anticipated life expectancy ≥20 weeks.

Key Exclusion Criteria:

1. Prior treatment with an agent that blocks the PD-1/PD-L1 pathway.
2. Prior treatment with other systemic immune-modulating agents as defined in the protocol
3. Major surgery or radiation therapy within 14 days of first administration of study drug
4. Has received treatment with an approved systemic therapy within 4 weeks of first dose of study drug, or has not yet recovered (ie, grade ≤1 or baseline) from any acute toxicities except for laboratory changes as described in the protocol
5. Has another malignancy that is progressing or requires active treatment and/or history of malignancy other than cervical cancer within 3 years of date of first planned dose of study drug as defined in the protocol
6. Has any condition that requires ongoing/continuous corticosteroid therapy (>10 mg prednisone/day or anti-inflammatory equivalent) within 4 weeks prior to the first dose of study drug. 7. Has ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments as defined in the protocol

NOTE: Other protocol-defined Inclusion/ Exclusion criteria apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2024-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (25):
- United States (2):
  - Arizona Oncology Associates, Tucson, Arizona
  - Regeneron Research Site, Orange, California
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent, East Flanders
  - UZ Leuven, Leuven, Vlaams Brabant
  - CHIREC Delta Hospital / Chirec Cancer Institute, Brussels
- Brazil (5):
  - Instituto Nacional de Cancer Jose Alencar Gomes da Silva ¿ INCA, Santo Cristo, Rio de Janeiro
  - Centro de Pesquisa em Oncologia - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro De Novos Tratamentos Itajai, Itajaí, Santa Catarina
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto COI de Pesquisa, Educacao e Gestao - COI Clinicas Barra Da Tijuca (COI Clinicas Oncologicas Integradas SA), Rio de Janeiro
- Italy (3):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) IRCCS, Meldola, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - IRCCS-Istituto Europeo di Oncologia, Milan
- Netherlands (4):
  - Maastricht University Medical Center, Maastricht, Limburg
  - University Medical Center Groningen, Groningen
  - Leiden Universitair Medisch Centrum (LUMC), Leiden
  - Radboudumc, Nijmegen
- State Budgetary Healthcare Institution Clinical Oncology Dispensary 1 Of Healthcare Department Of Krasnodar Region, Krasnodar, Krasnodarskiy Kray, Russia
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - University of Ulsan College of Medicine - Asan Medical Center (AMC), Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (3):
  - Hospital Doctor Josep Trueta - Institut Catala d'Oncologia (ICO), Girona, Catalonia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 229 participants were screened, and of these, 113 were enrolled and 116 were screen failures.
Groups:
- ISA 101b + Cemiplimab 350 mg Q3W: A dose of 100 μg/peptide ISA101b on days 1, 29, and 50 (total of 3 doses). Cemiplimab 350 mg (milligrams) given by IV (intravenous) infusion over 30 minutes Q3W (every 3 weeks) on days 8 and 29 in cycle 1, on days 1 and 22 in cycles 2 through 4, and on days 1, 22, and 43 in all subsequent cycles until disease progression or discontinuation of study drug
Period: Overall Study
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Started | 113
Completed | 0
Not Completed | 113
Not completed — Adverse Event | 1
Not completed — Progressive Disease | 71
Not completed — Death | 20
Not completed — Withdrawal by Subject | 12
Not completed — Sponsor Request | 9

BASELINE CHARACTERISTICS:
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 88
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 91
  More than one race | 2
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is determined by the proportion of participants with best overall response of complete response (CR) or partial response (PR) in the Full analysis set (FAS).
Time Frame: From enrollment to last dose (~up to 23 months)
Population: The full analysis set (FAS) included all enrolled participants who received any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Number analyzed (Participants) | 113
Percentage of Participants | 17.7 [10.7 to 24.7]

2. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: Treatment-emergent AEs (TEAEs) are defined as AEs that developed or worsened during the on-treatment period and treatment-related AEs that occur during post-treatment period.
Time Frame: From enrollment to last dose (~up to 23 months)
Population: The full analysis set (FAS) included all enrolled participants who received any study drug.
Measure: Number; unit: Events
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Number analyzed (Participants) | 113
Events | 877

3. Secondary Outcome: Number of Participants With Any Treatment Emergent Adverse Events (TEAEs)
Time Frame: From enrollment to last dose (~up to 23 months)
Population: The full analysis set (FAS) included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Number analyzed (Participants) | 113
Participants | 106

4. Secondary Outcome: Number of Participants With Any Treatment Emergent Adverse Events of Special Interest (TE AESIs)
Time Frame: From enrollment to last dose (~up to 23 months)
Population: The full analysis set (FAS) included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Number analyzed (Participants) | 113
Participants | 10

5. Secondary Outcome: Number of Participants With Any Serious TEAE
Time Frame: From enrollment to last dose (~up to 23 months)
Population: The full analysis set (FAS) included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Number analyzed (Participants) | 113
Participants | 31

6. Secondary Outcome: Number of Participants With at Least One Lab Abnormality
Time Frame: From enrollment to last dose (~up to 23 months)
Population: The full analysis set (FAS) included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Number analyzed (Participants) | 113
Participants
  Hematology Overall | 88
  Electrolytes Overall: number analyzed (Participants) | 104
  Electrolytes Overall | 56
  Liver function Overall: number analyzed (Participants) | 104
  Liver function Overall | 66
  Chemistry Overall: number analyzed (Participants) | 104
  Chemistry Overall | 33
  Coagulation Overall: number analyzed (Participants) | 98
  Coagulation Overall | 9

7. Secondary Outcome: Number of Participants With at Least One Lab Abnormality With Severity of ≥ Grade 3
Description: Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: From enrollment to last dose (~up to 23 months)
Population: The full analysis set (FAS) included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Number analyzed (Participants) | 113
Participants
  Hematology Overall | 27
  Electrolytes Overall: number analyzed (Participants) | 104
  Electrolytes Overall | 3
  Liver function Overall: number analyzed (Participants) | 104
  Liver function Overall | 3
  Chemistry Overall: number analyzed (Participants) | 104
  Chemistry Overall | 3
  Coagulation Overall: number analyzed (Participants) | 98
  Coagulation Overall | 0

8. Secondary Outcome: Duration of Response (DOR)
Time Frame: From enrollment to last dose (~up to 23 months)
Population: The full analysis set (FAS) included all enrolled participants who received any study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Number analyzed (Participants) | 113
months | 7.3 [3.5 to 19.9]

9. Secondary Outcome: Progression Free Survival (PFS)
Time Frame: From enrollment to last dose (~up to 23 months)
Population: The full analysis set (FAS) included all enrolled participants who received any study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Number analyzed (Participants) | 113
Months | 3.0 [1.7 to 4.0]

10. Secondary Outcome: Overall Survival (OS)
Time Frame: From enrollment to last dose (~up to 23 months)
Population: The full analysis set (FAS) included all enrolled participants who received any study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
Number analyzed (Participants) | 113
Months | 14.3 [11.7 to 17.3]

ADVERSE EVENTS:
Time Frame: From signing of informed consent to end of study (~up to 28 months)
Arm/Group | ISA 101b + Cemiplimab 350 mg Q3W
All-Cause Mortality (participants affected / at risk) | 68/113
Serious Adverse Events (participants affected / at risk) | 34/113
Other Adverse Events (participants affected / at risk) | 99/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISA 101b + Cemiplimab 350 mg Q3W (N=113)
Sepsis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Urosepsis (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Skin bacterial infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Renal haematoma (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urogenital fistula (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 (3)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (2)
Malaise (General disorders) | 1 (1)
Device dislocation (Product Issues) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (3)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISA 101b + Cemiplimab 350 mg Q3W (N=113)
Injection site reaction (General disorders) | 44 (58)
Pyrexia (General disorders) | 22 (32)
Fatigue (General disorders) | 21 (25)
Asthenia (General disorders) | 15 (16)
Oedema peripheral (General disorders) | 8 (8)
Influenza like illness (General disorders) | 7 (11)
Nausea (Gastrointestinal disorders) | 27 (35)
Vomiting (Gastrointestinal disorders) | 17 (22)
Abdominal pain (Gastrointestinal disorders) | 15 (16)
Constipation (Gastrointestinal disorders) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 16 (20)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 31 (51)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Hypothyroidism (Endocrine disorders) | 9 (9)
Hyperthyroidism (Endocrine disorders) | 9 (9)
Urinary tract infection (Infections and infestations) | 10 (13)
COVID-19 (Infections and infestations) | 6 (6)
Blood creatinine increased (Investigations) | 8 (11)
Aspartate aminotransferase increased (Investigations) | 7 (9)
Blood alkaline phosphatase increased (Investigations) | 7 (9)
Decreased appetite (Metabolism and nutrition disorders) | 14 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Headache (Nervous system disorders) | 12 (14)
Insomnia (Psychiatric disorders) | 8 (8)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (7)
Vaginal haemorrhage (Reproductive system and breast disorders) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8)
Hypotension (Vascular disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Alanine aminotransferase increased (Investigations) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the Sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT04646005/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT04646005/SAP_001.pdf